CLINICAL TRIAL: NCT02083458
Title: A New Infraclavicular Landmark-based Approach to the Axillary Vein as an Alternative Method of Central Venous Cannulation
Brief Title: An Infraclavicular Landmark-based Approach to the Axillary Vein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Ryszard Gawda, MD, Senior anesthesiologist, Uniwersytecki Szpital Kliniczny w Opolu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Axillary vein - WCM
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Critical Illness
Keywords: critical care; catheterization; axillary vein
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- axillary vein catheterization (Experimental): Catheterization of the axillary vein based on anatomical landmark.
  Interventions: Procedure: Catheterization of the axillary vein.

INTERVENTIONS:
Procedure: Catheterization of the axillary vein.

SUMMARY:
The central line placement is the widespread procedure performed in the intensive care and emergency medicine. Indications for this procedure are chiefly lack of peripheral catheters, administration some medications, renal replacement therapy, parenteral nutrition and hemodynamic monitoring.

The procedure is performed by percutaneous puncture of large vein of the neck and the thorax - internal jugular vein or subclavian vein, then insertion of guidewire through the needle and placement of the catheter over the guidewire. The tip of the catheter is situated in the superior vena cava.

There are two techniques of catheterizations: landmark-based and ultrasound-guided. The most frequently cannulated veins in landmark-based approach are internal jugular and subclavian vein. The cannulation of the axillary vein is not common procedure in the intensive care unit, mainly due its complicated original technique.

The primary intention of this study was to describe and assess usefulness and safety of the new landmark-based technique of catheterization of the axillary vein in patients admitted to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the intensive care unit with indications for central venous catheterization

Exclusion Criteria:

* chest wall deformities at the cannulations side
* major hemostasis disorders
* infections at the catheterization site
* age less than 18 years
* lack of patients consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Rate of successful catheterizations. | 24 hours
Procedure success rate depending on physician experience. | 24 hours

SECONDARY OUTCOMES:
Rate of early complications. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ryszard Gawda, MD, Principal Investigator — Department of Anesthesiology and Intensive Care, Publiczny Samodzielny Zaklad Opieki Zdrowotnej Wojewodzkie Centrum Medyczne w Opolu
Locations (1):
- Department of Anesthesiology and Intensive Care, Publiczny Samodzielny Zaklad Opieki Zdrowotnej Wojewodzkie Centrum Medyczne, Opole, Opole Voivodeship, Poland